CLINICAL TRIAL: NCT04398641
Title: Surgery for Deep Endometriosis of the Lower Rectum (Segmental/Disc) - a Prospective Comparison of Surgical Techniques Regarding Pre- and Postoperative Digestive Symptoms and Pain Outcomes
Brief Title: Surgery for Lower Rectum Deep Endometriosis (Segmental/Disc) - Prospective Comparison of Digestive Symptoms and Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Univ.-Doz. Dr.med.univ. Gernot Hudelist, MSc. (Other)
Responsible Party: Sponsor-Investigator, Univ.-Doz. Dr.med.univ. Gernot Hudelist, MSc., MD, MSc Clinical Lecturer, Woman and Health Private Clinic Vienna
Organization: Woman and Health Private Clinic Vienna (Other)
Other Study IDs: 2
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Endometriosis, Rectum
Keywords: Bowel endometriosis; Deep endometriosis (DE); Transanal disc excision (TADE); Nerve and vessel sparing segmental resection (NVSSR); Low Anterior Resection Syndrome (LARS); Digestive complaints; Gastrointestinal Quality of Life Index (GIQLI) by Eypasch
MeSH Terms: conditions — Endometriosis; Low Anterior Resection Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nerve and vessel sparing segmental resection (NVSSR): Women undergoing surgery for deep endometriosis of the lower rectum using the surgical technique of nerve and vessel sparing segmental resection (NVSSR)
  Interventions: Other: Evaluation of pre- and postoperative gastrointestinal functional outcomes
- Transanal disc excision (TADE): Women undergoing surgery for deep endometriosis of the lower rectum using the surgical technique of transanal disc excision (TADE)
  Interventions: Other: Evaluation of pre- and postoperative gastrointestinal functional outcomes

INTERVENTIONS:
Other: Evaluation of pre- and postoperative gastrointestinal functional outcomes — Gastrointestinal functional outcomes will be evaluated using the LARS and the GIQLI by Eypasch questionnaires.

SUMMARY:
Several studies show a significant drop in pain scores, improved fertility outcomes and amelioration of impaired sexual functioning in women following surgical resection of colorectal endometriosis. However, intermediate and long-term bowel dysfunction may occur as a consequence of radical surgery with typical symptoms such as constipation, feeling of incomplete evacuation, clustering of stools and urgency. This is described as low anterior resection syndrome (LARS).

The primary aim of this study is the prospective comparison of two surgical approaches for full thickness excision, i.e. transanal disc excision (TADE) and nerve-vessel sparing limited segmental resection (NVSSR), regarding gastrointestinal functional outcomes using the LARS / Gastrointestinal Quality of Life Index (GIQLI) by Eypasch questionnaires.

DETAILED DESCRIPTION:
Several studies show a significant drop in pain scores, improved fertility outcomes and amelioration of impaired sexual functioning in women following surgical resection of colorectal endometriosis. However, there is inceasing evidence that intermediate and long-term bowel dysfunction may occur as a consequence of radical surgery for rectal deep endometriosis (DE). Typical symptoms include constipation, feeling of incomplete evacuation, clustering of stools and urgency. This is described in the colorectal surgical literature as low anterior resection syndrome (LARS). The choice of operation is largely dependent on the extent of disease. Statistically significant differences in functional outcomes were found in favor of the conservative surgical approach, i.e. resection of endometriotic tissue with preservation of the luminal structure of the rectal wall thereby avoiding segmental bowel resection. In a recent retrospective multicentric cohort analysis, the incidence of LARS after either nerve and vessel sparing segmental resection (NVSSR) or transanal disc excision (TADE) performed for the surgical treatment of colorectal DE was assessed. All patients underwent a low rectum resection, with a resection line lower than 7cm from anal verge. In contrast to previoisly published data, no statistically significant difference between the incidence of the LARS among patients operated using TADE when compared to women treated by NVSSR were found. Interestingly, the occurence of LARS was positively associated with the use of protective ileo-or colostomy. A higher rate of severe complications was observed in the TADE group than among patients who underwent a NVSSR. Weaknesses of this study are the retrospective design and a possible bias in the TADE regarding larger DE nodules as well as the possibility of bowel dysfunction prior to surgery in women with DE.

The primary aim of the present study is the prospective comparison of two surgical approaches for full thickness excision of rectal DE resulting in an anastomotic height ≤7 cm distance from the anal verge. One technique involves the preservation of the residual luminal wall integrity (disc resection) known as Rouen technique/ TADE. The other technique involves limited resection of the bowel wall with preservation of all adjacent structures (autonomic pelvic plexus, rectal vascular supply) known as NVSSR. Gastrointestinal functional outcomes of the two procedures will be compared using the LARS / GIQLI by Eypasch questionnaires. Since digestive complaints may also be present presurgically, evaluation of digestive complaints will be recorded pre- and post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women undergoing full thickness excision of rectal deep endometriosis (DE) resulting in an anastomotic height ≤7 cm distance from the anal verge

Exclusion Criteria:

* Diagnosed or suspected malignancy
* Previous colorectal surgery
* Previous history of chronic inflammatory diseases of the gastrointestinal tract and/or chronic defecation dysfunction related to other factors such as birth trauma etc.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Premenopausal women undergoing full thickness excision of rectal deep endometriosis (DE) resulting in an anastomotic height ≤7 cm distance from the anal verge will be included in this study. These women will undergo either nerve and vessel sparing segmental resection (NVSSR) or transanal disc excision (TADE).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of gastrointestinal functional outcomes between groups using the LARS questionnaire | 4 to 24 months
  Gastrointestinal functional outcomes in the nerve and vessel sparing segmental resection (NVSSR) group versus the transanal disc excision (TADE) group will be compared using the Low Anterior Resection Syndrome (LARS) questionnaire.
  LARS questionnaire: scores range from a minimum of 0 to a maximum of 42 points; higher scores mean a worse outcome
Comparison of gastrointestinal functional outcomes between groups using the GIQLI by Eypasch questionnaire | 4 to 24 months
  Gastrointestinal functional outcomes in the nerve and vessel sparing segmental resection (NVSSR) group versus the transanal disc excision (TADE) group will be compared using the Gastrointestinal Quality of Life Index (GIQLI) by Eypasch questionnaire.
  GIQLI by Eypasch questionnaire: scores range from a minimum of 0 to a maximum of 144 points; higher scores mean a better outcome

SECONDARY OUTCOMES:
Prevalence of presurgical digestive complaints (LARS) | 1 day
  The prevalence of presurgical digestive complaints assessed using the LARS questionnaire will be evaluated.
Prevalence of presurgical digestive complaints (GIQLI by Eypasch) | 1 day
  The prevalence of presurgical digestive complaints assessed using the GIQLI by Eypasch questionnaire will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Gernot Hudelist, MD, MSc, Principal Investigator — Woman & Health Private Clinic Vienna
Locations (2):
- Austria (2):
  - Woman & Health Vienna, Vienna
  - Hospital St. John of God Vienna, Vienna